CLINICAL TRIAL: NCT01218893
Title: Immunization With Different Doses of Plasmodium Falciparum Sporozoites Under Chloroquine Prophylaxis
Acronym: ZonMw1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ZonMw1
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Plasmodium Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Immunization; Proguanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 15-15-15 (Active Comparator): This group will receive three times 15 infected mosquito bites under chloroquine prophylaxis, as we know that this dose is protective.
  Interventions: Drug: Chloroquine prophylaxis; Biological: Immunization; Biological: Plasmodium falciparum challenge; Drug: Malarone treatment
- 10-10-10 (Experimental): This group will receive three times 10 infected and 5 uninfected mosquito bites under chloroquine prophylaxis.
  Interventions: Drug: Chloroquine prophylaxis; Biological: Immunization; Biological: Plasmodium falciparum challenge; Drug: Malarone treatment
- 5-5-5 (Experimental): This group will receive three times 5 infected and 10 uninfected mosquitobites under chloroquine prophylaxis.
  Interventions: Drug: Chloroquine prophylaxis; Biological: Immunization; Biological: Plasmodium falciparum challenge; Drug: Malarone treatment
- 0-0-0 (Placebo Comparator): This group will receive three times 15 uninfected mosquitobites under prophylaxis.
  Interventions: Drug: Chloroquine prophylaxis; Biological: Immunization; Biological: Plasmodium falciparum challenge; Drug: Malarone treatment

INTERVENTIONS:
Drug: Chloroquine prophylaxis — The chloroquine dose used will be 300mg for the first two days, followed by 300mg per week, for 13 weeks.
Biological: Immunization — All groups will be immunised with mosquitobites. The number of infected mosquitoes differs per group, as clarified in group description.
Biological: Plasmodium falciparum challenge — Exposure to the bites of 5 Plasmodium falciparum infected mosquitoes.
Drug: Malarone treatment — When thick smear positive, of ar day 21 after challenge, all volunteers will be treated with malarone.
  Other Names: atovaquon/proguanil

SUMMARY:
Malaria is one of the major infectious diseases in the world with a tremendous impact on the quality of life significantly contributing to the ongoing poverty in endemic countries. It causes almost one million deaths per year, the majority of which are children under the age of five. The malaria parasite enters the human body through the skin, by the bite of an infected mosquito. Subsequently, it invades the liver and develops and multiplies inside the hepatocytes. After a week, the hepatocytes burst open and the parasites are released in the blood stream, causing the clinical phase of the disease.

As a unique opportunity to study malaria immunology and efficacy of immunisation strategies, a protocol has been developed in the past to conduct experimental human malaria infections (EHMIs). EHMIs generally involve small groups of malaria-naïve volunteers infected via the bites of P. falciparum infected laboratory-reared Anopheline mosquitoes. Although potentially serious or even lethal, P. falciparum malaria can be radically cured at the earliest stages of blood infection where risks of complications are virtually absent.

The investigators have shown previously that healthy human volunteers can be protected from a malaria mosquito (sporozoite) challenge by immunization with sporozoites (by mosquito bites) under chloroquine prophylaxis (CPS immunization). However, it is unknown how many mosquito bites are necessary to confer protection. Moreover, as all volunteers were protected in this study, no correlates of protection could be established. For future development of vaccines and understanding of protective immunity to malaria, it is important to investigate the lowest dose of CPS immunization that confers 100% protection and to find correlates of protection. Therefore, the present study aims to make the CPS immunization protocol more sensitive by lowering the number of infected mosquito bites, in order to study the underlying mechanisms of protection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 35 years healthy volunteers (males or females)
* Good health based on history and clinical examination
* Negative pregnancy test
* Use of adequate contraception for females
* All volunteers must sign the informed consent form demonstrating their understanding of the meaning and procedures of the study
* Volunteer agrees to inform the general practitioner and agrees to sign a request to release medical information concerning contra-indications for participation in the study
* Willingness to undergo a Pf mosquito challenge
* For volunteers not living in Leiden: agreement to stay in a hotel room close to the trial center during a part of the study (Day 5 after challenge till 3 days after treatment)
* Reachable (24/7) by mobile phone during the whole study period
* Living with a third party that could contact the clinicians in case of alteration of consciousness or agreement to stay in a hotel room close to the trial center during a part of the study (Day 5 after challenge till 3 days after treatment)
* Available to attend all study visits
* Agreement to refrain from blood donation to Sanquin or for other purposes, during the study period until 337.
* Willingness to undergo HIV, hepatitis B and hepatitis C tests
* Negative urine toxicology screening test at screening visit and day before challenge
* Willingness to take a prophylactic regime of chloroquine and curative regimen of Malarone®

Exclusion Criteria:

* History of malaria
* Plans to travel to malaria endemic areas during the study period
* Plans to travel outside of the Netherlands during the challenge period
* Previous participation in any malaria vaccine study and/or positive serology for Pf
* Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
* History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
* History of arrhythmias or prolonged QT-interval
* Positive family history in 1st and 2nd degree relatives for cardiac disease < 50 years old
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system
* Clinically significant abnormalities in electrocardiogram (ECG) at screening
* Body Mass Index (BMI) below 18 or above 30 kg/m2
* Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis
* Positive HIV, HBV or HCV tests
* Participation in any other clinical study within 30 days prior to the onset of the study
* Enrollment in any other clinical study during the study period
* Pregnant or lactating women
* Volunteers unable to give written informed consent
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study
* A history of psychiatric disease
* Known hypersensitivity to Malarone® or chloroquine
* The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months of study onset (inhaled and topical corticosteroids are allowed) and during the study period
* Contra-indications to Malarone® or chloroquine including treatment taken by the volunteer that interferes with Malarone® or chloroquine
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including asplenia
* Co-workers of the departments of Medical Microbiology, Parasitology, or Internal Medicine of the Leiden University medical Centre
* A history of sickle cell anemia, sickle cell trait, thalassemia, thalassemia trait or G6PD deficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Period to thick smear positivity after challenge in groups 1, 2, 3 and 4 | 21 days after challenge (day 218 of study)
Parasitemia and kinetics of parasitemia as measured by PCR in groups 1, 2, 3 and 4 | 21 days after challenge (day 218 of study)
Frequency of signs or symptoms in groups 1, 2, 3 and 4 | Day 21 after challenge (day 218 of study)

SECONDARY OUTCOMES:
Cellular immune response between groups 1, 2, 3 and 4 | Day 0 - day 337 of study
Antibody production between groups 1, 2, 3 and 4 | Day 0 - day 337 of study
Cytokine profile in groups 1, 2, 3 and 4 | Day 0 - day 337 of study

CONTACTS AND LOCATIONS:
Overall Officials: Leo G Visser, MD, PhD, Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, Netherlands

REFERENCES:
- [Derived] Nahrendorf W, Scholzen A, Bijker EM, Teirlinck AC, Bastiaens GJ, Schats R, Hermsen CC, Visser LG, Langhorne J, Sauerwein RW. Memory B-cell and antibody responses induced by Plasmodium falciparum sporozoite immunization. J Infect Dis. 2014 Dec 15;210(12):1981-90. doi: 10.1093/infdis/jiu354. Epub 2014 Jun 25. PMID 24970846
- [Derived] Bijker EM, Teirlinck AC, Schats R, van Gemert GJ, van de Vegte-Bolmer M, van Lieshout L, IntHout J, Hermsen CC, Scholzen A, Visser LG, Sauerwein RW. Cytotoxic markers associate with protection against malaria in human volunteers immunized with Plasmodium falciparum sporozoites. J Infect Dis. 2014 Nov 15;210(10):1605-15. doi: 10.1093/infdis/jiu293. Epub 2014 May 27. PMID 24872326